CLINICAL TRIAL: NCT04766658
Title: Gargle Phonation in Individuals With Muscle Tension Dysphonia
Brief Title: A Study to Evaluate Effects of Gargle Phonation in Voice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Diana M. Orbelo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20-004267
Record Dates: First submitted 2021-01-29; First posted 2021-02-23 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Voice Disorders; Muscle Tension Dysphonia; Speech Therapy
MeSH Terms: conditions — Voice Disorders; Communication Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water Swallow Intervention First (Other): Subjects will complete voice recordings after water swallows and then perform voice recordings after gargle phonation.
  Interventions: Other: Water swallow
- Gargle Phonation Intervention First (Other): Subjects will complete voice recordings after gargle phonation and then perform voice recordings after gargle phonation.
  Interventions: Other: Gargle Phonation

INTERVENTIONS:
Other: Gargle Phonation — Subjects will gargle water while making sound
  Arms: Gargle Phonation Intervention First
Other: Water swallow — Subjects will hold water in their mouth for 5 seconds and swallow
  Arms: Water Swallow Intervention First

SUMMARY:
The purpose of this study is to assess subjects with muscle tension dysphonia for perceived effort and acoustic effects of gargle phonation compared to baseline and a sham water swallow.

DETAILED DESCRIPTION:
This study assesses perceived effort following baseline talking, water swallows and gargle phonation. In addition to perceived effort, acoustic and perceptual analyses will be conducted on the recorded voice samples using vowel sounds, the Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) and Hearing in Noise Sentences (HINT).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a primary or secondary muscle tension dysphonia based clinical assessment with a Mayo clinic speech language pathologist or other Mayo Clinic otolaryngology care provider in Rochester or Phoenix/Scottsdale locations.
* Age 18 through 89.
* Able to provide informed consent.

Exclusion Criteria:

* Anyone not meeting inclusion criteria.
* Anyone unable or unwilling to provide informed consent.
* Anyone unable to complete questionnaires or participate in voice recording.
* Anyone with severe neurological voice or speech disorders.
* Moderate or severe dysphagia for thin liquids.
* Non-English speakers (English as a second language may be included).
* Extensive laryngeal surgery or other surgery or medical condition that may significantly alter the motor or sensory aspects of the larynx.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Rating of Effort Baseline | Baseline
  Measured using patient self-reported Borg effort scale where 0=no vocal effort and 10=maximum vocal effort.
Rating of Effort Post Swallow | After water swallow intervention, approximately 5 minutes
  Measured using patient self-reported Borg effort scale where 0=no vocal effort and 10=maximum vocal effort.
Rating of Effort Post Gargle | After gargle phonation intervention, approximately 5 minutes
  Measured using patient self-reported Borg effort scale where 0=no vocal effort and 10=maximum vocal effort.

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Orbelo, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials